CLINICAL TRIAL: NCT06663800
Title: Additional Effects of Ujjayi Pranayama on Pulmonary Function in Post Coronary Artery Bypass Graft
Brief Title: Additional Effects of Ujjayi Pranayama
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MSPT0193 Kulsoom
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Function; Coronary Artery Disease
Keywords: Ujjayi Paranyama; Coronary artery bypass grafting; Pulmonary Function
MeSH Terms: conditions — Coronary Artery Disease | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm:1 Pranayama (Experimental): Arm:1 Additional effects of Ujjayi Pranayama
  Interventions: Other: Ujjayi Paranayama
- arm: 2 (standard protocol) (Other): Arm:2 (standard protocol)
  Interventions: Other: Standard Protocol

INTERVENTIONS:
Other: Ujjayi Paranayama — Inhale or breathe in slowly while taking a deep, prolonged breath through both nostrils. As you inhale, attempt to tighten your throat and feel the air in your throat. Air should not come into contact with the interior of the nose. When air enters the throat, an odd sound is made. Allow the breath to be loose and easy while you slightly tighten the back of your throat and hiss lightly as you breathe in and out. The sound isn't forced, but it should be loud enough for someone to hear you if they were close. Now close your right nostril and release the breath through your left. As you exhale, try making the sound HHHHHAAAA
  Arms: arm:1 Pranayama
Other: Standard Protocol — Control Group will perform Deep Breathing Adhering to a FITT model protocol, with a frequency of 5 days. Intensity set at 8 repetitions, duration range from 10 to 15 minutes
  Arms: arm: 2 (standard protocol)

SUMMARY:
Studying the impact of Ujjayi pranayama on post-Coronary Artery Bypass Grafting (CABG) patients has the potential to positively influence healthcare. This research fosters a patient-centered approach, enhancing cardio respiratory function. Patient education on these practices can empower individuals, actively contributing to their recovery and overall well-being.

DETAILED DESCRIPTION:
. Exercises such as Ujjayi pranayama lower heart rate and benefit high blood pressure sufferers. To determine additional effects of Ujjayi pranayama on pulmonary function in post coronary artery bypass Graft (CABG).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have 1st post op Day
* Hemodynamically stable & well oriented patient
* Extubated Patient
* Voluntary based patients
* After approval of surgeon CABG patient were recruited
* Tachypnea

Exclusion Criteria:

* Hemodynamically unstable,
* Uncontrolled Hypertension,
* MSK disease,
* Any previous history of tuberculosis,
* Neurological disease ,
* Acute exacerbation of COAD & Asthma Attack,
* Any trauma, anxiety or Rib fracture case ,
* During surgery complaint of graft failure ,
* Unwilling to participate ,
* Postural Hypotension.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Borg dyspnea | 5days
  (Modified CR-10 is used to assess the degree of dyspnea, rated from 0 to 10. Zero means nothing at all, 0.5=extremely slight, 1=very slight, 2=slight, 3=moderate, 4=somewhat severe, 5=severe, 7=very severe, 9=extremely severe (almost maximal)
PFT | 5days
  Spirometer is simple test used to help diagnose and monitor certain lung conditions by measuring how much air you can breathe out in one forced breathe. Which is a small machine attached by a cable to a mouthpiece. This spirometer yielded generally reproducible results that were generally valid compared to laboratory-based spirometry. The use of this handheld spirometer in clinical, occupational, and research settings seems justified

SECONDARY OUTCOMES:
Cardiac monitors | 5days
  After 5, 10, 15, 20, and 30 minutes of pranayama in the study group and without pranayama in the control group, recordings of HR, SBP, DBP, RR, SpO2

CONTACTS AND LOCATIONS:
Overall Officials: Maria Razzaq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Railway general hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
maintaining confidentiality